CLINICAL TRIAL: NCT02116790
Title: Study of the Efficacy of Co-administration of an NSAID With a Dopamine Agonist in the Alleviation of Acute Cutaneous Inflammatory Pain in Healthy Subjects
Brief Title: Efficacy of Co-administration of an NSAID With a Dopamine Agonist In Healthy Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00083465; R01DE022746 (NIH)
Record Dates: First submitted 2014-02-17; First posted 2014-04-17 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Acute Pain
Keywords: acute; pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Naproxen; carbidopa, levodopa drug combination; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Group (Placebo Comparator): 10 participants will be given two pills: both will be placebos
  Interventions: Drug: Placebo
- Standard Treatment / Positive Control Group (Active Comparator): 10 participants will be given two pills: both will be Naproxen (each pill = 250mg, total dose = 500mg)
  Interventions: Drug: Naproxen
- Experimental Group #1 (Active Comparator): 10 participants will be given two pills: one will be Naproxen (250 mg) and the other will be of Sinemet (carbidopa/levodopa 12.5mg/50mg)
  Interventions: Drug: Naproxen; Drug: Sinemet
- Experimental Group #2 (Active Comparator): 10 participants will be given two pills: one will be Naproxen (250 mg) and the other will be of Sinemet (carbidopa/levodopa 25mg/100mg )
  Interventions: Drug: Naproxen; Drug: Sinemet

INTERVENTIONS:
Drug: Naproxen — Subjects will take one 250mg Naproxen capsule
  Other Names: Aleve; Anaprox; Antalgin; Apranax; Feminax Ultra; Flanax; Inza; Midol Extended Relief; Nalgesin; Naposin; Naprelan; Naprogesic; Naprosyn; Narocin; Proxen; Soproxen; Synflex; Xenobid
  Arms: Experimental Group #1; Experimental Group #2; Standard Treatment / Positive Control Group
Drug: Sinemet — Subjects will take one 12.5mg/50mg Sinemet.
  Other Names: Carbidopa/levodopa; Levocarb; Pharmacopa; Atamet; Apo-Levocarb; Co-careldopa
  Arms: Experimental Group #1
Drug: Sinemet — Subjects will take one 25mg/100mg Sinemet.
  Other Names: Carbidopa/levodopa; Levocarb; Pharmacopa; Atamet; Apo-Levocarb; Co-careldopa
  Arms: Experimental Group #2
Drug: Placebo — Subjects will take two placebos.
  Other Names: Sugar Pill
  Arms: Control Group

SUMMARY:
Findings from the investigator's lab and others' show the involvement of the brain's mesolimbic circuitry in pain perception and evaluation, as well as during the transition from acute to chronic pain states in both humans and animals. Dopamine (DA) is one of the main neurotransmitters in this circuitry, and it is possible it could have an intimate role in pain processing, chronicity, and related anatomical and functional neuroplasticity. In this study, the investigators first need to know if the combination of l-dopa and Naproxen is safe and efficacious in humans with acute pain, and if so, at what doses. For the present study, healthy pain-free participants will be injected with a small bolus of capsaicin subcutaneously to induce acute cutaneous inflammatory pain. Capsaicin is ideal for this study because it causes a characteristic inflammatory response that is almost always accompanied with pain, has a well-validated dose-response curve, and has effects that will go away completely in a few hours after administration, causing no permanent damage to study subjects. Effects of capsaicin will be measured by changes (decreases) from baseline in thermal and tactile thresholds, as well as by verbally reported cutaneous pain levels (on a scale from 0-10). Participants will also be given study medication in the form of a placebo, one drug, or a combination of drugs before capsaicin injection to allow for any analgesic effects to peak before pain onset. For those receiving active medication, they will either receive Naproxen with placebo or the combination of naproxen and l-dopa (the latter of which will be in one of two different doses). This will allow the investigators to investigate (1) whether co-administration of naproxen and l-dopa has analgesic effects in low levels of acute pain in humans, (2) if this combination is pain-alleviating, whether it is equally as or more efficacious than naproxen, which is the clinical standard of treatment, and finally (3) what dose provides the most analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Must be currently healthy and have none of the exclusion criteria listed below.
* Must be at least 18 years of age.
* Must be able to communicate (speak and write) in English.
* Must demonstrate that they understand what the study entails and requires of them.
* Must be able to dedicate the amount of time (~3 hours) to participate in the study.

Exclusion Criteria:

* History of chronic pain of any kind
* Have a current episode of acute pain of any kind (including stomach ache, headache, muscle ache, etc)
* History of psychiatric illness or brain injury
* History of substance abuse
* History of motor impairments
* History of another chronic disease (such as heart disease, celiac's, bronchial asthma, etc)
* Have a diagnosis of narrow-angle glaucoma
* History or presence of high blood pressure
* History or presence of melanoma cancer
* Currently on a high-protein diet
* Women who are pregnant, trying to get pregnant, or breastfeeding
* Known or suspected allergies to capsaicin, peppers, levodopa, carbidopa, naproxen, NSAIDs, rubbing alcohol (in the medical wipes), or lidocaine
* History or presence of dermatological disorder, including contact dermatitis and a history of skin allergies in general
* Presence of a skin lesion in the areas to be tested

Prohibited Medication:

* Aliskiren
* ACE inhibitors
* Angiotensin 2 receptor blockers
* Cidofovir
* Corticosteroids
* Anti-platelet drugs
* Blood-thinners
* Another NSAID
* MAOIs
* Tetrabenazine
* Anti-depressants
* Anti-psychotics
* Metoclopramide
* Phenytoin
* Papaverine
* Sedatives or muscle relaxers
* Tryptan/L-tryptophan
* DA agonists/antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
VAS pain scale | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Apkar V Apkarian, PhD, Principal Investigator — Northwestern University